CLINICAL TRIAL: NCT05288686
Title: Use of Superparamagnetic Iron Oxide (SPIO) Versus Conventional Radioisotope and Patent Blue Dye in Sentinel Lymph Node Detection for Breast Cancer: a Randomized Controlled Trial
Brief Title: Use of Superparamagnetic Iron Oxide (SPIO) in Sentinel Lymph Node Detection for Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, MAN Chi Mei Vivian, Honorary Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKUCTR-2709
Record Dates: First submitted 2022-03-10; First posted 2022-03-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Sentinel Lymph Node
Keywords: superparamagnetic iron oxide; sentinel lymph node detection rate
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Masking Description: Masking is not possible due to the different color of the injected tracer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIO arm (Experimental): Superparamagnetic iron oxide guided sentinel lymph node mapping
  Interventions: Procedure: sentinel lymph node biopsy procedure
- Control arm (Active Comparator): Conventional radioisotope and blue dye guided sentinel lymph node mapping
  Interventions: Procedure: sentinel lymph node biopsy procedure

INTERVENTIONS:
Procedure: sentinel lymph node biopsy procedure — Patient received respective tracer injection and sentinel lymph node biopsy was performed in the operation theatre with the corresponding device.

SUMMARY:
Sentinel lymph node biopsy is mandatory during breast cancer operation for disease staging and treatment. The localization of sentinel lymph node is by the injection of radioisotope and blue dye, which is the gold standard. However the use of radioisotope and blue dye are associated with specific drawbacks. Superparamagnetic iron oxide is a magnetic tracer which is FDA-approved for sentinel lymph node localization. The hypothesis of this study is superparamagnetic iron oxide can replace the conventional dual mapping of radioisotope and blue dye in the detection of sentinel lymph nodes for early breast cancers.

DETAILED DESCRIPTION:
Sentinel lymph node biopsy has replaced axillary dissection as the standard of care in clinically node negative breast cancer. Lymphatic mapping with radioisotope and blue dye were most studied tracer agents and their combination was shown to give the highest nodal identification rate and lowest false negative rate. However the use of radioisotope is strictly monitored due to its radioactivity and blue dye is associated with potential allergic reactions and skin tattoo. Superparamagnetic iron oxide is non-radioactive. It gives an audible signal with the magnetometer and a brown color as visual cue. It has demonstrated comparable nodal identification rate with the conventional method in multiple non-inferiority trials in Europe and the USA. There was no randomized controlled trial for a head-to-head comparison between these mapping technique. The hypothesis of this study is superparamagnetic iron oxide alone can replace the conventional dual mapping of radioisotope and blue dye.

Previous literature suggested the nodal detection rate for conventional method and SPIO was around 97%. Assuming a non-inferiorly limit of 5%, with a power of 80% and 5% significance level, the number of patients per treatment arm should be 144. We will need a sample size of 300 patients, taking into account a loss to follow-up of <5%.

All patients recruited will be provided full explanation of the study and written voluntary consents will be obtained before randomization.

All data will be prospectively collected by dedicated research assistant and computerized into a database. All statistical analysis will be performed with Statistical Product and Service Solution (SPSS) version 24. Missing information will be marked and significant missing data will be excluded from analysis. Chi-square test will be used to compare discrete variables and student T test or Mann Whitney U test for continuous variables. P value less than 0.05 will be considered statistically significant.

Personal data will be obtained by principal investigator and dedicated research assistant to allow analysis of the results. These data will be anonymous, only identified by the first three letters of patient's name. The file will be encrypted and stored in the study institution. All the information will be solely for research purpose and kept strictly confidential.

Research subjects will be provided with phone contacts for any questions or emergency related to the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients with clinical T1-3N0 invasive ductal carcinoma or invasive lobular carcinoma planned for breast conservative surgery or mastectomy, with sentinel lymph node biopsy
* Patients planned for upfront operation or neoadjuvant chemotherapy are allowed

Exclusion Criteria:

* Patients with hypersensitivity to dextran compounds, iron or blue dye
* Patients with iron overload disease
* Pregnant or lactating patients
* Patients with pacemaker or other implantable metallic devices in chest wall or prosthesis in shoulder
* Mentally incompetent patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
sentinel lymph node detection rate per patient | At the time of operation
  Successful sentinel lymph node localization for each arm

SECONDARY OUTCOMES:
Number of sentinel lymph nodes detected | At the time of operation
  Number of sentinel lymph nodes detected in each arm
Duration of sentinel lymph node biopsy | Duration of the operation from incision of axillary fascia to satisfactory nodal basin count
  Duration of sentinel lymph node biopsy procedure in each arm
Detection rate of pathologically involved sentinel lymph nodes | At operation
  Detection rate of malignant sentinel lymph nodes in each arm
Duration of skin stain | post-operative 3 month, 6 month, 12 month and 18 month
  Duration of blue stain (from blue dye) and brown stain (from SPIO) in respective arm

CONTACTS AND LOCATIONS:
Overall Officials: Ava Kwong, Professor, Study Director — university
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Douek M, Klaase J, Monypenny I, Kothari A, Zechmeister K, Brown D, Wyld L, Drew P, Garmo H, Agbaje O, Pankhurst Q, Anninga B, Grootendorst M, Ten Haken B, Hall-Craggs MA, Purushotham A, Pinder S; SentiMAG Trialists Group. Sentinel node biopsy using a magnetic tracer versus standard technique: the SentiMAG Multicentre Trial. Ann Surg Oncol. 2014 Apr;21(4):1237-45. doi: 10.1245/s10434-013-3379-6. Epub 2013 Dec 10. PMID 24322530
- [Result] Thill M, Kurylcio A, Welter R, van Haasteren V, Grosse B, Berclaz G, Polkowski W, Hauser N. The Central-European SentiMag study: sentinel lymph node biopsy with superparamagnetic iron oxide (SPIO) vs. radioisotope. Breast. 2014 Apr;23(2):175-9. doi: 10.1016/j.breast.2014.01.004. Epub 2014 Jan 29. PMID 24484967
- [Result] Pinero-Madrona A, Torro-Richart JA, de Leon-Carrillo JM, de Castro-Parga G, Navarro-Cecilia J, Dominguez-Cunchillos F, Roman-Santamaria JM, Fuster-Diana C, Pardo-Garcia R; Grupo de Estudios Senologicos de la Sociedad Espanola de Patologia Mamaria (SESPM). Superparamagnetic iron oxide as a tracer for sentinel node biopsy in breast cancer: A comparative non-inferiority study. Eur J Surg Oncol. 2015 Aug;41(8):991-7. doi: 10.1016/j.ejso.2015.04.017. Epub 2015 May 12. PMID 25997792
- [Result] Rubio IT, Diaz-Botero S, Esgueva A, Rodriguez R, Cortadellas T, Cordoba O, Espinosa-Bravo M. The superparamagnetic iron oxide is equivalent to the Tc99 radiotracer method for identifying the sentinel lymph node in breast cancer. Eur J Surg Oncol. 2015 Jan;41(1):46-51. doi: 10.1016/j.ejso.2014.11.006. Epub 2014 Nov 15. PMID 25466980
- [Result] Houpeau JL, Chauvet MP, Guillemin F, Bendavid-Athias C, Charitansky H, Kramar A, Giard S. Sentinel lymph node identification using superparamagnetic iron oxide particles versus radioisotope: The French Sentimag feasibility trial. J Surg Oncol. 2016 Apr;113(5):501-7. doi: 10.1002/jso.24164. Epub 2016 Jan 12. PMID 26754343
- [Result] Ghilli M, Carretta E, Di Filippo F, Battaglia C, Fustaino L, Galanou I, Di Filippo S, Rucci P, Fantini MP, Roncella M. The superparamagnetic iron oxide tracer: a valid alternative in sentinel node biopsy for breast cancer treatment. Eur J Cancer Care (Engl). 2017 Jul;26(4). doi: 10.1111/ecc.12385. Epub 2015 Sep 14. PMID 26365441
- [Result] Karakatsanis A, Christiansen PM, Fischer L, Hedin C, Pistioli L, Sund M, Rasmussen NR, Jornsgard H, Tegnelius D, Eriksson S, Daskalakis K, Warnberg F, Markopoulos CJ, Bergkvist L. The Nordic SentiMag trial: a comparison of super paramagnetic iron oxide (SPIO) nanoparticles versus Tc(99) and patent blue in the detection of sentinel node (SN) in patients with breast cancer and a meta-analysis of earlier studies. Breast Cancer Res Treat. 2016 Jun;157(2):281-294. doi: 10.1007/s10549-016-3809-9. Epub 2016 Apr 27. PMID 27117158
- [Derived] Chiu HY, Man V, Suen D, Kwong A. Skin-Staining From Superparamagnetic Iron Oxide (SPIO) for Sentinel Lymph Node Sampling-Follow-Up Results From a Randomized Trial. World J Surg. 2026 Jan;50(1):21-28. doi: 10.1002/wjs.70173. Epub 2025 Nov 22. PMID 41273311